CLINICAL TRIAL: NCT04368572
Title: Comparison of the Efficacy of Hypnosis on Pain and Anxiety Versus Standard Care During Lumbar Puncture for Etiological Diagnosis of Cognitive Impairment
Brief Title: Efficacy of Hypnosis on Pain and Anxiety During Lumbar Puncture for Etiological Diagnosis of Cognitive Impairment
Acronym: POESY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-A00447-50
Record Dates: First submitted 2020-04-17; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Cognitive Impairment; Alzheimer's Disease
Keywords: Hypnosis; Lumbar puncture; Cognitive impairment; Alzheimer's Disease; Cerebrospinal fluid
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: the investigator will blindly collect the subject's self-rated pain and anxiety scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumbar puncture under hypnosis (Experimental): Hypnosis is the only act added by protocol to patients receiving a lumbar puncture as part of the etiological assessment of cognitive disorders
  Interventions: Behavioral: Hypnosis
- lumbar puncture without hypnosis (Active Comparator): Lumbar puncture is performed by a physician assisted by a nurse or a psychologist who reassure the patient during the installation and the procedure.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — An interview assesses the patient's level of anxiety, interests and dissociative abilities. Hypnosis is done by following the steps:
  First step: reception and installation of the patient Second step: induction phase Third step: hypnotic trance phase Fourth step: reorientation phase

SUMMARY:
Lumbar puncture is a diagnostic procedure performed as part of the etiological assessment of cognitive disorders. Despite good tolerance and very rare complications, lumbar puncture is still perceived as being painful or anxiety-provoking by patients. Hypnosis could improve pain and anxiety when performing lumbar puncture.

DETAILED DESCRIPTION:
Lumbar puncture is an invasive procedure potentially inducing pain and anxiety indicated in elderly patients for cognitive assessment. Indeed, the measure of amyloid biomarkers and tau in the cerebrospinal fluid is useful in the etiological diagnosis of cognitive disorders. With the ageing of the population and the increase incidence of cognitive disorders, this diagnostic procedure will be more and more frequent. Many studies have shown the efficiency of hypnosis during invasive procedure, especially in young children. The absence of side-effect is a major asset in elderly patients at high iatrogenic risk. It represents an interesting alternative to anxiolytic or sedative treatments. Nevertheless, its effectiveness in the elderly during lumbar puncture remains to be demonstrated. Investigators hypothesized that hypnosis may decrease pain and anxiety during lumbar puncture associated to setting comfort situation (relational care, music, transcutaneous anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years old
* Indication for a lumbar puncture for etiological diagnosis of cognitive impairment
* Understanding French Language
* Written and informed consent for this study signed by the patient
* Affiliated to Health Insurance

Exclusion Criteria:

* MMS< 17 or cognitive impairment not allowing informed consent
* Contraindication to lumbar puncture
* Refusal to sign the written and informed consent
* Patient deprived of freedom by court or administrative order

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain during the lumbar puncture | 1 day
  Pain is assessed by visual analogue scale, a self-reported pain rating scale (0 "no pain" to 10 "worst pain")

SECONDARY OUTCOMES:
Pain assessed by the physician during the lumbar puncture using Algoplus© score | 1 day
  Algoplus© score is an acute pain-behaviour scale for older people with inability to communicate verbally (0 "No pain" to 30 "worst pain")
Assessment of anxiety during the lumbar puncture according a visual analogue scale | 1 day
  Anxiety is evaluated by the patient with a visual analogue scale (0 "No anxiety" to 10 "Worst anxiety)
Assessment of anxiety during the lumbar puncture according a numeric scale | 1 day
  Anxiety is evaluated by the physician with a numeric scale (0 "No anxiety" to 10 "Worst anxiety)
Assessment of anxiety during the lumbar puncture by monitoring the heart rate | 1 day
Assessment of anxiety during the lumbar punctureby monitoring the Galvanic Skin Response | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Lilamand, MD, Study Chair — Geriatric Department, Bichat hospital
Locations (1):
- Geriatric Department, Bichat hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Courtois-Amiot P, Cloppet-Fontaine A, Poissonnet A, Benit E, Dauzet M, Raynaud-Simon A, Paquet C, Lilamand M. Hypnosis for pain and anxiety management in cognitively impaired older adults undergoing scheduled lumbar punctures: a randomized controlled pilot study. Alzheimers Res Ther. 2022 Sep 2;14(1):120. doi: 10.1186/s13195-022-01065-w. PMID 36056417